CLINICAL TRIAL: NCT00911989
Title: Endoscopic Visualization During a Laparoscopic Sleeve Gastrectomy Procedure
Brief Title: Laparoscopic Sleeve Gastrectomy With Endoscopic Visualization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-08-0008
Record Dates: First submitted 2009-05-31; First posted 2009-06-03 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Morbid Obesity
Keywords: Obesity; Weight Loss
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Transvaginal Sleeve Gastrectomy (Other): Transvaginal Sleeve Gastrectomy using Steerable Flex Trocar (SFT) for transvaginal endoscope placement (endoscopic visualization)
  Interventions: Device: NOTES toolbox

INTERVENTIONS:
Device: NOTES toolbox — Using SFT for endoscope access during Transvaginal Sleeve Gastrectomy procedure. Visualization will occur through endoscope

SUMMARY:
The main objective of this trial is to evaluate endoscopic visualization during a laparoscopic sleeve gastrectomy (LSG) procedure using an endoscope inserted transvaginally through a new device called a Steerable Flex Trocar (SFT).

ELIGIBILITY:
Inclusion Criteria

Women will be enrolled in this study who:

* Are willing to give consent and comply with evaluation and treatment schedule;
* Are 21 to 60 years of age (inclusive), post menopausal, or otherwise no longer expect to bear children, e.g., previous tubal ligation;
* Are a candidate for surgical weight loss intervention (meets ASMBS and NIH criteria);
* Have no significant psychopathology that could limit the subject's ability to understand the procedure, comply with medical, surgical, and/or behavioral recommendations;
* Agree to refrain from any type of elective procedures that would affect body weight such as abdominal lipoplasty or liposuction, mammoplasty, or removal of excess skin for the duration of the trial;
* Are American Society of Anesthesiologists (ASA) Class I, II, or III); and
* Have a negative pregnancy test (for women of childbearing potential).

Exclusion Criteria

Subjects will be excluded from the study for any of the following:

* Previous pelvic surgery other than transverse C-sections and/or tubal ligation;
* Enlarged uterus;
* Evidence of pelvic malignancy on a screening ultrasound;
* Documented history of drug and/or alcohol abuse within 2 years of the Screening Visit;
* Previous malabsorptive or restrictive procedures performed for the treatment of obesity;
* Unable or unwilling to attend follow-up visits and examinations;
* Planned or predicted concurrent surgical procedure;
* Any medical condition which precludes compliance with the study;
* Immunocompromised such as that resulting from chronic oral steroid use, chemotherapeutic agents, or immune deficiency disorders;
* Conditions that, in the opinion of the investigator, may jeopardize the subject's well-being and/or the soundness of this clinical study;
* History or presence of pre-existing autoimmune connective tissue disease, e.g., systemic lupus erythematosus or scleroderma;
* Use of prescription or over the counter weight reduction medications or supplements, participation in weight-loss programs, or change in smoking habits within 8 weeks of the Screening Visit and for the duration of study participation;
* Participation in another clinical trial within 8 weeks of the Screening Visit and for the duration of this trial (unless previously approved by the investigator and Sponsor); or
* Any condition which precludes compliance with the study (investigator discretion).

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Myers, MD, FACS, Principal Investigator — Riverside Methodist Hospital
Locations (1):
- Riverside Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Transvaginal Sleeve Gastrectomy
Started | 4
Completed | 3
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Transvaginal Sleeve Gastrectomy
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48.3 (11.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Procedures Completed With Successful Endoscopic Visualization.
Description: The goal of the study was to evaluate the feasibility of endoscopic visualization during a laparoscopic sleeve gastrectomy procedure using an endoscope inserted transvaginally through a steerable flex trocar. The number of subjects in whom the procedure was completed with endoscopic visualization was recorded.
Time Frame: Assessed intra-operatively
Population: All subjects on whom the surgery was attempted represent the primary analysis population.
Measure: Number; unit: participants
Groups:
- Transvaginal Sleeve Gastrectomy: All subjects on whom the surgery was attempted.
Arm/Group | Transvaginal Sleeve Gastrectomy
Number analyzed (Participants) | 4
participants | 4

ADVERSE EVENTS:
Time Frame: Adverse events collected from informed consent date to 12 months post surgery.
Arm/Group | Transvaginal Sleeve Gastrectomy
Serious Adverse Events (participants affected / at risk) | 1/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transvaginal Sleeve Gastrectomy (N=4)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Transvaginal Sleeve Gastrectomy (N=4)
Abnormal faeces (Gastrointestinal disorders) | 1 (1)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4)
Oesophageal pain (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1)
Post procedural complications (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Procedural nausea (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (4)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less